CLINICAL TRIAL: NCT01592006
Title: A Pilot Study on the Efficicay and Safety of Pegylated Interferon, Ribavirin and Telaprevir in Recurrent Hepatitis C Virus (HCV) Infection in Orthotopic Liver Transplant (OLT) Recipients.
Brief Title: Pegylated Interferon, Ribavirin, Telaprevir in Hepatitis C Virus Infection in Orthotopic Liver Transplant Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0156
Record Dates: First submitted 2012-04-27; First posted 2012-05-04 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C
Keywords: hepatitis C virus; liver transplant recipient
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCV, LT, Pegasys, ribavirin, telaprevir (Experimental): Patients are being asked to be part of this arm because they are orthotopic liver transplant recipients (OLT) and have the Hepatitis C Virus (HCV). They will be given the study drugs Pegasys, ribavirin and telaprevir
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: telaprevir

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Patients will be treated with pegylated interferon alfa-2a (Pegasys®) 180 mcg SQ per week for 12 weeks, followed by pegylated interferon alfa-2a (Pegasys®) and ribavirin for another 36 weeks. Patients will be assessed at periodic intervals for safety and adverse effects. Following completion of therapy, patients will be followed for another 24 weeks to determine sustained response.
Drug: Ribavirin — Patients will be given ribavirin 600-1200 mg PO per day for 12 weeks, followed by pegylated interferon alfa-2a (Pegasys®) and ribavirin for another 36 weeks. Patients will be assessed at periodic intervals for safety and adverse effects. Following completion of therapy, patients will be followed for another 24 weeks to determine sustained response.
Drug: telaprevir — Patients will be given telaprevir 750 mg tid (Incivek®) for 12 weeks, followed by pegylated interferon alfa-2a (Pegasys®) and ribavirin for another 36 weeks. Patients will be assessed at periodic intervals for safety and adverse effects. Following completion of therapy, patients will be followed for another 24 weeks to determine sustained response.

SUMMARY:
Patients are being asked to be part of this study because they are a liver transplant recipient and have the Hepatitis C Virus (HCV). Current routine treatment for HCV for liver transplant patients includes taking two medications called pegylated interferon alfa-2a (Pegasys®) and ribavirin. Patients Pegasys and ribavirin are FDA approved for the treatment of HCV.

This study will evaluate the safety and efficacy of adding a third drug called telaprevir for the experimental treatment of HCV in liver transplant patients. The combination of Pegasys, ribavirin and telaprevir is currently FDA approved for the treatment of HCV, but is specifically not FDA approved for HCV patients who have had a liver transplant. This is because more information is needed about possible drug interactions between telaprevir and cyclosporine, or telaprevir and tacrolimus-based immunosuppressive drugs, which are typically part of routine care for transplant patients.

Studies have shown that the addition of telaprevir greatly increases the efficacy of Pegasys and ribavirin for the treatment of HCV. However, these studies did not include adequate information on transplant patients due to the potential drug interactions.

The investigators hope to gather more information about the safety and efficacy of telaprevir given in combination with Pegasys and ribavirin in the liver transplant patients who have HCV that is not well controlled with Pegasys and ribavirin alone.

DETAILED DESCRIPTION:
BACKGROUND:

Cirrhosis from HCV is the most common indication for OLT. Unfortunately, disease recurrence in the allograft is virtually universal. The spectrum of disease recurrence ranges from minimal inflammation to severe cholestasis as well as cirrhosis, leading to allograft failure. Previous reports indicated a comparable survival rate between patients who received OLT for HCV and those who received OLT for other indications. More recent data, however, suggested that HCV-positive recipients have significantly impaired patient and allograft survival following OLT as compared to HCV-negative recipients. Approximately 20% of patients with recurrent HCV have cirrhosis at 5 years post-OLT.

Attempts to treat HCV recurrence in OLT recipients have had limited success. Sustained virologic responses (SVR) have only been seen in up to 30% of patients with genotype 1 infection, whereas SVR has been higher at 42-46% for non-transplant counterparts. Most recently, the addition of telaprevir to pegylated interferon and ribavirin to comprise the triple therapy in the nontransplant HCV-infected population has led to significantly higher sustained virologic response rate (SVR) of 75% when compared to 44% observed in the control arm which received pegylated interferon and ribavirin. Its side effect profile was acceptable to allow the FDA to approve the drug on May 23, 2011. However, there is no data on the efficacy and safety of telaprevir in OLT recipients. In fact, its use in this population is greatly hindered by a significant drug-drug interaction with the major immunosuppressive agents used in OLT, namely tacrolimus and cyclosporine. Telaprevir increases cyslosporine exposure by 4.6 fold and its half-life by 3.5 fold. It increases tacrolimus exposure to 70 fold and its half-life by 4.9 fold. Clearly, the doses of these immunosuppressive agents need to be adjusted at the start and end of telaprevir therapy.

The primary aim of our study is to determine the safety and efficacy of pegylated interferon alfa-2a (Pegasys®), ribavirin, and telaprevir therapy in liver transplant recipients with hepatitis C recurrence who are maintained on cyclosporine or tacrolimus-based immunosuppression. We hypothesize that triple therapy will have better sustained virologic response rates than the current standard of care, pegylated interferon and ribavirin, with an acceptable side-effect profile.

STUDY DESIGN:

Prospective, open-label, single center pilot study. All patients will receive the study drug along with the standard regimen of pegylated interferon and ribavirin.

DRUG DOSE AND TREATMENT DURATION:

Patients will be treated with pegylated interferon alfa-2a (Pegasys®) 180 mcg SQ per week, ribavirin 800-1200 mg PO per day (weight-based) for 48 weeks. Telaprevir 750 mg PO tid will be administered for the first 12 weeks. Following completion of therapy, patients will be followed for another 24 weeks to determine sustained response.

*Doses lower than 800 mg/day may be used by the investigator in patients with renal insufficiency (as ribavirin is renally excreted), at the investigator's discretion.

RESEARCH PROTOCOL:

This prospective study will include patients who have histologic evidence of recurrent HCV infection who are maintained on cyclosporine-based immunosuppression.

Patients who qualify for the study will be identified from the Liver Transplant Clinic. Patients will be treated with pegylated interferon alfa-2a (Pegasys®) 180 mcg SQ per week, ribavirin 600-1200 mg PO per day, and telaprevir 750 mg tid (Incivek®) for 12 weeks, followed by pegylated interferon alfa-2a (Pegasys®) and ribavirin for another 36 weeks. Patients will be assessed at periodic intervals for safety and adverse effects as delineated in the Schedule of Assessments (Appendix A). Growth factors such as erythropoietin and filgastrim will be allowed in the event that signficiant anemia and thrombocytopenia develops during therapy, at the discretion of the investigator.

The HCV RNA will be measured at baseline and weeks 2, 4, 8, 12, 24, 36 and 48 of therapy as well as during follow-up. Response to therapy is defined by HCV RNA <1000 IU/ml at weeks 4, 8, and 12 of therapy, which will allow continuation of treatment. Telaprevir will be discontinued if HCV RNA is >1000 IU/ml at weeks 4 or 8 of therapy, and pegylated interferon and ribavirin will be discontinued if HCV RNA is still detectable by week 24 of therapy.

Cyclosporine or tacrolimus trough levels will be drawn at baseline, days 1,2, 3, 4,5, 8, and to be continued every 2-3 days. The cyclosporine or tacrolimus dose will be cut by 50% at baseline and cyclosporine or tacrolimus dose adjustments will be made to maintain the level within the targeted therapeutic range. Once two consecutive levels within the targeted therapeutic range have been achieved, levels will be drawn weekly for the first month then biweekly until the end of telaprevir treatment. After the last dose of telaprevir, cyclosporine or tacrolimus levels will be drawn on days 1, 3, 5, 7 and to be continued every other day, and cyclosporine or tacrolimus dose adjustments will be made to maintain the level within the targeted therapeutic range. Once two consecutive levels within the targeted therapeutic range have been achieved, levels will be drawn in a week and then monthly for up to week 24 of therapy. Patients who complete therapy will continue to be followed for 24 weeks to determine their sustained virologic response.

STATISTICAL ANALYSIS:

This is a pilot, single arm study that evaluates the efficacy and safety of triple therapy in recurrent HCV. All clinical and laboratory data will be entered into a computer database. Categorical variables will be expressed as proportions and continuous variables will be expressed in mean values.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age.
* Detectable plasma HCV-RNA by qualitative PCR assay.
* HCV genotype 1 infection,
* Documented recurrent hepatitis C by liver biopsy within the past year.
* On cyclosporine or tacrolimus-based immunosuppression
* Negative urine pregnancy test before initiating the treatment for women of childbearing potential.
* Willingness of the patient and all potentially childbearing partners to use a reliable form of effective contraception during the study, unless the patient or partner is surgically sterile or post-menopausal.
* Willingness to undergo provide informed consent and comply with study requirements.

Exclusion Criteria:

* Genotype non-1 HCV infection.
* Women who are pregnant or breast-feeding.
* Male partners of women who are pregnant.
* Evidence of co-infection with HIV or hepatitis B.
* History of severe psychiatric disease.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, lupus erythematosus, rheumatoid arthritis, etc.)
* History of clinically significant pulmonary disease.
* History of severe cardiac disease.
* History of malignancy where risk of recurrence is >20% within 2 years.
* History of uncontrolled seizure disorder.
* History of poorly controlled thyroid disease.
* History of poorly controlled diabetes mellitus.
* History of severe retinopathy.
* Active gout.
* History or evidence of severe medical illness that, in the opinion of the investigator, makes the patient unsuitable for pegylated interferon alfa-2a treatment (Pegasys®).
* Inability or unwillingness to abstain from alcohol throughout the entire study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Te, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since new better drug options had became available, the intervention drug of this study was no longer the best option for the patients. Thus this study was terminated.
Groups:
- HCV, LT, Pegasys, Ribavirin, Telaprevir: Patients will be treated with Pegylated interferon alfa-2a (Pegasys®) 180 mcg SQ per week, Ribavirin 800-1200 mg PO per day (weight-based) for 48 weeks. Telaprevir 750 mg PO tid will be administered for the first 12 weeks. Following completion of therapy, patients will be followed for another 24 weeks to determine sustained response.
Period: Overall Study
Arm/Group | HCV, LT, Pegasys, Ribavirin, Telaprevir
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HCV, LT, Pegasys, Ribavirin, Telaprevir
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Triple Antiviral Therapy
Description: To evaluate the efficacy of triple antiviral therapy, consisting of pegylated interferon alfa-2a (Pegasys®), ribavirin, and telaprevir therapy in liver transplant recipients with hepatitis C. This will be measured and reported by sustained virologic response (defined as undetectable HCV RNA in the blood 24 weeks after completing therapy [SVR24])
Time Frame: 3 years from start of study
Measure: Number; unit: percentage of participants
Arm/Group | HCV, LT, Pegasys, Ribavirin, Telaprevir
Number analyzed (Participants) | 3
percentage of participants | 100

2. Secondary Outcome: Safety of Triple Antiviral Therapy in HCV Infected OLT Recipients
Description: Tolerability and Safety will be measured and reported by serious adverse events.
Time Frame: 6 years from the start of the study
Measure: Number; unit: participants
Arm/Group | HCV, LT, Pegasys, Ribavirin, Telaprevir
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HCV, LT, Pegasys, Ribavirin, Telaprevir
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HCV, LT, Pegasys, Ribavirin, Telaprevir (N=3)
Anorectal discomfort (Gastrointestinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 3
Irritable (Psychiatric disorders) | 2
MVA (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Headache (Nervous system disorders) | 2
Mouth sores (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes